CLINICAL TRIAL: NCT04051320
Title: Characterizing the Neural Substrates of Irritability in Women: an Experimental Neuroendocrine Model
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 19-0401; R21MH119615-01 (NIH)
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Results first posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-05

CONDITIONS: Perinatal Depression; Post Partum Depression; Depression, Postpartum; Depression
Keywords: Irritability; Estrogen; Progesterone; Lupron Depot; Mood Disorders; Perinatal Depression; Postpartum; Hormones; Physiological effects of drugs; Reproductive Control Agents; Mental Disorders; Hormone Intervention; Functional Magnetic Resonance Imaging
MeSH Terms: conditions — Depression, Postpartum; Depression; Mood Disorders; Mental Disorders | interventions — Leuprolide; Estradiol; Tablets; Progesterone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hormone Sensitive Women (HS+) (Experimental): Participants will take leuprolide acetate (lupron) via intramuscular injection, for 2 months. Participants will take 2 mg of estradiol twice daily and 200 mg of progesterone twice daily for 2 weeks.
  Interventions: Drug: Leuprolide Acetate 3.75 MG/ML; Drug: Estradiol 2 Mg tablet; Drug: Micronized progesterone
- Hormone Insensitive Women (HS-) (Experimental): Participants will take leuprolide acetate (lupron) via intramuscular injection, for 2 months. Participants will take 2 mg of estradiol twice daily and 200 mg of progesterone twice daily for 2 weeks.
  Interventions: Drug: Leuprolide Acetate 3.75 MG/ML; Drug: Estradiol 2 Mg tablet; Drug: Micronized progesterone

INTERVENTIONS:
Drug: Leuprolide Acetate 3.75 MG/ML — 3.75 mg/month leuprolide acetate intramuscular injection
  Other Names: Lupron
Drug: Estradiol 2 Mg tablet — 2 mg estradiol tablet
  Other Names: Estrace
Drug: Micronized progesterone — 200 mg micronized progesterone tablets
  Other Names: Prometrium

SUMMARY:
The proposed study involves experimentally manipulating reproductive hormones in nonpregnant, euthymic women to create a scaled down version of the changes that occur during pregnancy and the postpartum period. This endocrine manipulation paradigm, which the investigators have shown provokes irritability in past studies, will be used to examine the neurocircuitry underlying irritability under baseline and hormone challenge conditions among women who are hormone sensitive (HS+; n=15) and non-hormone sensitive (HS-; n=15). The long-term goal of this research is to advance understanding of the neural systems underlying both the triggering of and susceptibility to irritability in women. The objective of the current project is to examine whether HS+ show differences in the behavioral activation system relative to HS- under baseline and hormone challenge conditions using functional magnetic resonance imaging (fMRI) and behavioral tests.

DETAILED DESCRIPTION:
Irritability, defined as a predisposition to exhibit anger, is a prominent, defining symptom of perinatal depression (PND) and many other neuropsychiatric disorders. Despite the near ubiquity of irritability across disorders, the neural dysfunction underlying the vulnerability to, onset of, and exacerbation of irritability is understudied and poorly understood. The proposed study involves experimentally manipulating reproductive hormones in nonpregnant, euthymic women to create a scaled down version of the changes that occur during pregnancy and the postpartum period. This endocrine manipulation paradigm, which the investigators have shown provokes irritability in past studies, will be used to examine the neurocircuitry underlying irritability under baseline and hormone challenge conditions among women who are hormone sensitive (HS+; n=15) and non-hormone sensitive (HS-; n=15). The long-term goal of this research is to advance understanding of the neural systems underlying both the triggering of and susceptibility to irritability in women. The objective of the current project is to examine whether HS+ show differences in the behavioral activation system relative to HS- under baseline and hormone challenge conditions using functional magnetic resonance imaging (fMRI) and behavioral tests. The investigator's central hypothesis is that reproductive hormone changes are associated with dysregulated threat and reward processing and consequent irritability in HS+. The rationale for the proposed study is that employing a scaled down model of puerperal hormonal events permits the identification of a group of individuals homogeneous for hormone sensitivity (HS+), hence creating the best opportunity for disentangling the specific changes in brain function due to reproductive hormones (i.e., HS-) from those accompanying reproductive hormone-precipitated affective dysfunction (i.e., HS+). Because women will act as their own controls across time, this study design also allows for a powerful evaluation of state and trait variables that may contribute to irritability, including both threat and reward processing. Identifying both state and trait markers of irritability, and disentangling them from the effects of reproductive hormones on brain and behavior, will allow for the identification of neural substrates of irritability susceptibility that can be investigated across neuropsychiatric disorders. The expected outcome of this research is the identification of neural circuits underlying both the susceptibility to and mediation of irritability.

ELIGIBILITY:
Inclusion Criteria:

Participants will include healthy, euthymic 22-45 year old women with a history of postpartum depression (n=15) and women without such a history (n=15). Thus, only participants capable of giving informed consent will be enrolled. Participants will be compensated upon completion of the study.

Inclusion Criteria. Group 1: Women with a history of perinatal depression

* A history of a the Diagnostic Statistic Manual of Mental Disorders - fifth edition (DSM-V) major depression episode that occurred within 6 weeks of childbirth (as determined by a SCID interview) and remitted at least one year prior to enrollment in the study;
* has been well for a minimum of one year;
* a regular menstrual cycle for at least three months;
* age 22-45;
* medication free (including birth control pills);.

Group 2: Healthy Controls

* Controls will meet all inclusion criteria specified above except they must not have any past or present Axis I diagnosis or evidence of menstrually related mood disorders.

A structured clinical interview for DSM-V (SCID) will be administered to all women prior to study entry. Any woman with a current axis I psychiatric diagnosis will be excluded from participating in this protocol.

Exclusion Criteria:

Patients will not be permitted to enter this protocol if they have important clinical or laboratory abnormalities including any of the following:

* current axis I psychiatric diagnosis (based on a structured clinical interview for DSM-V (SCID);
* endometriosis;
* undiagnosed enlargement of the ovaries;
* liver disease;
* breast cancer;
* a history of blood clots in the legs or lungs;
* undiagnosed vaginal bleeding;
* porphyria;
* diabetes mellitus;
* malignant melanoma;
* gallbladder or pancreatic disease;
* heart or kidney disease;
* cerebrovascular disease (stroke);
* cigarette smoking;
* a history of suicide attempts or psychotic episodes requiring hospitalization;
* recurrent migraine with aura;
* pregnancy-related medical conditions such as hyperemesis gravidarum, preeclampsia and toxemia, deep vein thrombosis (DVT) and bleeding diathesis;
* Any woman with a first degree relative (immediate family) with premenopausal breast cancer or breast cancer presenting in both breasts or any woman who has multiple family members (greater than three relatives) with postmenopausal breast cancer will also be excluded from participating in this protocol;

Any woman meeting the Stages of Reproductive Aging Workshop Criteria (STRAW) for perimenopause will be excluded from participation. Specifically, the investigators will exclude any woman with an elevated plasma follicle stimulating hormone (FSH) level (> 14 IU/L) and with menstrual cycle variability of > 7 days different from their normal cycle length.

Pregnant women will be excluded from participation (patients will be warned not to become pregnant during the study and will be advised to employ barrier contraceptive methods), and women who become pregnant (although unlikely because of the hormone manipulation) will be withdrawn. The use of leuprolide acetate is not recommended during pregnancy. Prior to treatment, a complete physical, including a serum β-human chorionic gonadotropin (HCG) test for pregnancy. Participants will be seen at the outpatient clinic on a regular biweekly basis. All participants will be required to use non-hormonal forms of birth control (e.g., barrier methods) to avoid pregnancy during this study. Participants will also undergo urine toxicology and pregnancy tests on the day of each of the two fMRI scans. If a woman becomes pregnant during the study, she will not complete the fMRI scan, and the hormone protocol will be discontinued.

Ages: 22 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Men will not be included in this study, given the stated purpose of studying irritability in women with and without perinatal depression.
Enrollment: 23 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Crystal E Schiller, PhD, Principal Investigator — UNC Dept of Psychiatry
Locations (1):
- University of North Carolina at Chapel Hill School of Medicine, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 18 to 24 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: SAP, Analytic Code
Time Frame: Deidentified individual data that supports the results will be shared beginning 18 to 24 months following publication.
Access Criteria: Approval from an IRB, IEC, or REB, as applicable and execution of a data use/sharing agreement with UNC.

REFERENCES:
- [Background] Vidal-Ribas P, Brotman MA, Valdivieso I, Leibenluft E, Stringaris A. The Status of Irritability in Psychiatry: A Conceptual and Quantitative Review. J Am Acad Child Adolesc Psychiatry. 2016 Jul;55(7):556-70. doi: 10.1016/j.jaac.2016.04.014. Epub 2016 May 6. PMID 27343883
- [Background] Battle DE. Diagnostic and Statistical Manual of Mental Disorders (DSM). Codas. 2013;25(2):191-2. doi: 10.1590/s2317-17822013000200017. No abstract available. PMID 24413388
- [Background] Fava M, Hwang I, Rush AJ, Sampson N, Walters EE, Kessler RC. The importance of irritability as a symptom of major depressive disorder: results from the National Comorbidity Survey Replication. Mol Psychiatry. 2010 Aug;15(8):856-67. doi: 10.1038/mp.2009.20. Epub 2009 Mar 10. PMID 19274052
- [Background] Perlis RH, Fraguas R, Fava M, Trivedi MH, Luther JF, Wisniewski SR, Rush AJ. Prevalence and clinical correlates of irritability in major depressive disorder: a preliminary report from the Sequenced Treatment Alternatives to Relieve Depression study. J Clin Psychiatry. 2005 Feb;66(2):159-66; quiz 147, 273-4. PMID 15705000
- [Background] Leibenluft E, Cohen P, Gorrindo T, Brook JS, Pine DS. Chronic versus episodic irritability in youth: a community-based, longitudinal study of clinical and diagnostic associations. J Child Adolesc Psychopharmacol. 2006 Aug;16(4):456-66. doi: 10.1089/cap.2006.16.456. PMID 16958570
- [Background] Price M, van Stolk-Cooke K. Examination of the interrelations between the factors of PTSD, major depression, and generalized anxiety disorder in a heterogeneous trauma-exposed sample using DSM 5 criteria. J Affect Disord. 2015 Nov 1;186:149-55. doi: 10.1016/j.jad.2015.06.012. Epub 2015 Jul 29. PMID 26241663
- [Background] Van Voorhees EE, Dennis PA, Elbogen EB, Fuemmeler B, Neal LC, Calhoun PS, Beckham JC. Characterizing anger-related affect in individuals with posttraumatic stress disorder using ecological momentary assessment. Psychiatry Res. 2018 Mar;261:274-280. doi: 10.1016/j.psychres.2017.12.080. Epub 2018 Jan 3. PMID 29329048
- [Background] Penn DL, Spaulding W, Reed D, Sullivan M. The relationship of social cognition to ward behavior in chronic schizophrenia. Schizophr Res. 1996 Jul 5;20(3):327-35. doi: 10.1016/0920-9964(96)00010-2. PMID 8827860
- [Background] Bilgi MM, Taspinar S, Aksoy B, Oguz K, Coburn K, Gonul AS. The relationship between childhood trauma, emotion recognition, and irritability in schizophrenia patients. Psychiatry Res. 2017 May;251:90-96. doi: 10.1016/j.psychres.2017.01.091. Epub 2017 Feb 3. PMID 28192770
- [Background] McGuire K, Fung LK, Hagopian L, Vasa RA, Mahajan R, Bernal P, Silberman AE, Wolfe A, Coury DL, Hardan AY, Veenstra-VanderWeele J, Whitaker AH. Irritability and Problem Behavior in Autism Spectrum Disorder: A Practice Pathway for Pediatric Primary Care. Pediatrics. 2016 Feb;137 Suppl 2:S136-48. doi: 10.1542/peds.2015-2851L. Epub 2016 Feb 1. PMID 26908469
- [Background] Alper KR, Barry JJ, Balabanov AJ. Treatment of psychosis, aggression, and irritability in patients with epilepsy. Epilepsy Behav. 2002 Oct;3(5S):13-18. doi: 10.1016/s1525-5069(02)00500-5. PMID 12609315
- [Background] Lopez OL, Becker JT, Sweet RA, Klunk W, Kaufer DI, Saxton J, Habeych M, DeKosky ST. Psychiatric symptoms vary with the severity of dementia in probable Alzheimer's disease. J Neuropsychiatry Clin Neurosci. 2003 Summer;15(3):346-53. doi: 10.1176/jnp.15.3.346. PMID 12928511
- [Background] Scott LN, Stepp SD, Hallquist MN, Whalen DJ, Wright AGC, Pilkonis PA. Daily shame and hostile irritability in adolescent girls with borderline personality disorder symptoms. Personal Disord. 2015 Jan;6(1):53-63. doi: 10.1037/per0000107. PMID 25580673
- [Background] Leibenluft E. Pediatric Irritability: A Systems Neuroscience Approach. Trends Cogn Sci. 2017 Apr;21(4):277-289. doi: 10.1016/j.tics.2017.02.002. Epub 2017 Mar 6. PMID 28274677
- [Background] Williamson JA, O'Hara MW, Stuart S, Hart KJ, Watson D. Assessment of postpartum depressive symptoms: the importance of somatic symptoms and irritability. Assessment. 2015 Jun;22(3):309-18. doi: 10.1177/1073191114544357. Epub 2014 Jul 24. PMID 25059681
- [Background] Schiller CE, Johnson SL, Abate AC, Schmidt PJ, Rubinow DR. Reproductive Steroid Regulation of Mood and Behavior. Compr Physiol. 2016 Jun 13;6(3):1135-60. doi: 10.1002/cphy.c150014. PMID 27347888
- [Background] Postpartum Depression: Action Towards Causes and Treatment (PACT) Consortium. Heterogeneity of postpartum depression: a latent class analysis. Lancet Psychiatry. 2015 Jan;2(1):59-67. doi: 10.1016/S2215-0366(14)00055-8. Epub 2015 Jan 8. PMID 26359613
- [Background] Bloch M, Schmidt PJ, Danaceau M, Murphy J, Nieman L, Rubinow DR. Effects of gonadal steroids in women with a history of postpartum depression. Am J Psychiatry. 2000 Jun;157(6):924-30. doi: 10.1176/appi.ajp.157.6.924. PMID 10831472
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Salum GA, Mogg K, Bradley BP, Stringaris A, Gadelha A, Pan PM, Rohde LA, Polanczyk GV, Manfro GG, Pine DS, Leibenluft E. Association between irritability and bias in attention orienting to threat in children and adolescents. J Child Psychol Psychiatry. 2017 May;58(5):595-602. doi: 10.1111/jcpp.12659. Epub 2016 Oct 26. PMID 27782299
- [Background] Blair RJ. The Neurobiology of Impulsive Aggression. J Child Adolesc Psychopharmacol. 2016 Feb;26(1):4-9. doi: 10.1089/cap.2015.0088. Epub 2015 Oct 14. PMID 26465707
- [Background] Stringaris A, Cohen P, Pine DS, Leibenluft E. Adult outcomes of youth irritability: a 20-year prospective community-based study. Am J Psychiatry. 2009 Sep;166(9):1048-54. doi: 10.1176/appi.ajp.2009.08121849. Epub 2009 Jul 1. PMID 19570932
- [Background] Savage J, Verhulst B, Copeland W, Althoff RR, Lichtenstein P, Roberson-Nay R. A genetically informed study of the longitudinal relation between irritability and anxious/depressed symptoms. J Am Acad Child Adolesc Psychiatry. 2015 May;54(5):377-84. doi: 10.1016/j.jaac.2015.02.010. Epub 2015 Feb 28. PMID 25901774
- [Background] Stoddard J, Tseng WL, Kim P, Chen G, Yi J, Donahue L, Brotman MA, Towbin KE, Pine DS, Leibenluft E. Association of Irritability and Anxiety With the Neural Mechanisms of Implicit Face Emotion Processing in Youths With Psychopathology. JAMA Psychiatry. 2017 Jan 1;74(1):95-103. doi: 10.1001/jamapsychiatry.2016.3282. PMID 27902832
- [Background] Brotman MA, Kircanski K, Stringaris A, Pine DS, Leibenluft E. Irritability in Youths: A Translational Model. Am J Psychiatry. 2017 Jun 1;174(6):520-532. doi: 10.1176/appi.ajp.2016.16070839. Epub 2017 Jan 20. PMID 28103715
- [Background] Deveney CM, Connolly ME, Haring CT, Bones BL, Reynolds RC, Kim P, Pine DS, Leibenluft E. Neural mechanisms of frustration in chronically irritable children. Am J Psychiatry. 2013 Oct;170(10):1186-94. doi: 10.1176/appi.ajp.2013.12070917. PMID 23732841
- [Background] Vitaro F, Barker ED, Boivin M, Brendgen M, Tremblay RE. Do early difficult temperament and harsh parenting differentially predict reactive and proactive aggression? J Abnorm Child Psychol. 2006 Oct;34(5):685-95. doi: 10.1007/s10802-006-9055-6. Epub 2006 Oct 18. PMID 17048109
- [Background] Gray, J. A. The Psychology of Fear and Stress. (CUP Archive, 1987).
- [Background] McNaughton N, Corr PJ. A two-dimensional neuropsychology of defense: fear/anxiety and defensive distance. Neurosci Biobehav Rev. 2004 May;28(3):285-305. doi: 10.1016/j.neubiorev.2004.03.005. PMID 15225972
- [Background] Cox EQ, Raines C, Kimmel M, Richardson E, Stuebe A, Meltzer-Brody S. Comprehensive Integrated Care Model to Improve Maternal Mental Health. J Obstet Gynecol Neonatal Nurs. 2017 Nov-Dec;46(6):923-930. doi: 10.1016/j.jogn.2017.08.003. Epub 2017 Sep 6. PMID 28888920
- [Background] Spinelli MG, Endicott J, Goetz RR, Segre LS. Reanalysis of efficacy of interpersonal psychotherapy for antepartum depression versus parenting education program: initial severity of depression as a predictor of treatment outcome. J Clin Psychiatry. 2016 Apr;77(4):535-40. doi: 10.4088/JCP.15m09787. PMID 27137422
- [Background] Forty L, Jones L, Macgregor S, Caesar S, Cooper C, Hough A, Dean L, Dave S, Farmer A, McGuffin P, Brewster S, Craddock N, Jones I. Familiality of postpartum depression in unipolar disorder: results of a family study. Am J Psychiatry. 2006 Sep;163(9):1549-53. doi: 10.1176/ajp.2006.163.9.1549. PMID 16946179
- [Background] First, M. B., Spitzer, R. L., Gibbon, M. & Williams, J. B. W. Structured Clinical Interview for DSM-IV-TR Axis I Disorders, Research Version, Non-patient Edition. (SCID-I/NP). (Biometrics Research, New York State Psychiatric Institute, 2002).
- [Background] Clark, L. A. Schedule for Nonadaptive and Adaptive Personality (SNAP). (University of Minnesota Press, 1993).
- [Background] Endicott J, Nee J, Cohen J, Halbreich U. Premenstrual changes: patterns and correlates of daily ratings. J Affect Disord. 1986 Mar-Apr;10(2):127-35. doi: 10.1016/0165-0327(86)90035-2. PMID 2941469
- [Background] Watson D, O'Hara MW, Simms LJ, Kotov R, Chmielewski M, McDade-Montez EA, Gamez W, Stuart S. Development and validation of the Inventory of Depression and Anxiety Symptoms (IDAS). Psychol Assess. 2007 Sep;19(3):253-68. doi: 10.1037/1040-3590.19.3.253. PMID 17845118
- [Background] Carver, C. S. & White, T. L. Behavioral Inhibition, Behavioral Activation, and Affective Responses to Impending Reward and Punishment: The Bis/bas Scales. J. Pers. Soc. Psychol. 67, 319-333 (1994).
- [Background] Wright, K. A., Lam, D. H. & Brown, R. G. Reduced approach motivation following nonreward: Extension of the BIS/BAS scales. Personal. Individ. Differ. 47, 753-757 (2009).
- [Background] Beaver JD, Lawrence AD, van Ditzhuijzen J, Davis MH, Woods A, Calder AJ. Individual differences in reward drive predict neural responses to images of food. J Neurosci. 2006 May 10;26(19):5160-6. doi: 10.1523/JNEUROSCI.0350-06.2006. PMID 16687507
- [Background] Simon JJ, Walther S, Fiebach CJ, Friederich HC, Stippich C, Weisbrod M, Kaiser S. Neural reward processing is modulated by approach- and avoidance-related personality traits. Neuroimage. 2010 Jan 15;49(2):1868-74. doi: 10.1016/j.neuroimage.2009.09.016. Epub 2009 Sep 18. PMID 19770056
- [Background] Tseng WL, Moroney E, Machlin L, Roberson-Nay R, Hettema JM, Carney D, Stoddard J, Towbin KA, Pine DS, Leibenluft E, Brotman MA. Test-retest reliability and validity of a frustration paradigm and irritability measures. J Affect Disord. 2017 Apr 1;212:38-45. doi: 10.1016/j.jad.2017.01.024. Epub 2017 Jan 23. PMID 28135689
- [Background] Rich BA, Schmajuk M, Perez-Edgar KE, Pine DS, Fox NA, Leibenluft E. The impact of reward, punishment, and frustration on attention in pediatric bipolar disorder. Biol Psychiatry. 2005 Oct 1;58(7):532-9. doi: 10.1016/j.biopsych.2005.01.006. Epub 2005 Jun 13. PMID 15953589
- [Background] Rich BA, Schmajuk M, Perez-Edgar KE, Fox NA, Pine DS, Leibenluft E. Different psychophysiological and behavioral responses elicited by frustration in pediatric bipolar disorder and severe mood dysregulation. Am J Psychiatry. 2007 Feb;164(2):309-17. doi: 10.1176/ajp.2007.164.2.309. PMID 17267795
- [Background] Rich BA, Holroyd T, Carver FW, Onelio LM, Mendoza JK, Cornwell BR, Fox NA, Pine DS, Coppola R, Leibenluft E. A preliminary study of the neural mechanisms of frustration in pediatric bipolar disorder using magnetoencephalography. Depress Anxiety. 2010 Mar;27(3):276-86. doi: 10.1002/da.20649. PMID 20037920
- [Background] Mogg, K. & Bradley, B. P. Attentional Bias in Generalized Anxiety Disorder Versus Depressive Disorder. Cogn. Ther. Res. 29, 29-45 (2005).
- [Background] Bradley BP, Mogg K, White J, Groom C, de Bono J. Attentional bias for emotional faces in generalized anxiety disorder. Br J Clin Psychol. 1999 Sep;38(3):267-78. doi: 10.1348/014466599162845. PMID 10532148
- [Background] Mogg K, Bradley BP. Some methodological issues in assessing attentional biases for threatening faces in anxiety: a replication study using a modified version of the probe detection task. Behav Res Ther. 1999 Jun;37(6):595-604. doi: 10.1016/s0005-7967(98)00158-2. PMID 10372472
- [Background] Golomb BA, Cortez-Perez M, Jaworski BA, Mednick S, Dimsdale J. Point subtraction aggression paradigm: validity of a brief schedule of use. Violence Vict. 2007;22(1):95-103. doi: 10.1891/vv-v22i1a006. PMID 17390565
- [Background] Dougherty DM, Bjork JM, Huckabee HC, Moeller FG, Swann AC. Laboratory measures of aggression and impulsivity in women with borderline personality disorder. Psychiatry Res. 1999 Mar 22;85(3):315-26. doi: 10.1016/s0165-1781(99)00011-6. PMID 10333383
- [Background] Hooley JM, Gruber SA, Scott LA, Hiller JB, Yurgelun-Todd DA. Activation in dorsolateral prefrontal cortex in response to maternal criticism and praise in recovered depressed and healthy control participants. Biol Psychiatry. 2005 Apr 1;57(7):809-12. doi: 10.1016/j.biopsych.2005.01.012. PMID 15820239
- [Background] Grimm S, Beck J, Schuepbach D, Hell D, Boesiger P, Bermpohl F, Niehaus L, Boeker H, Northoff G. Imbalance between left and right dorsolateral prefrontal cortex in major depression is linked to negative emotional judgment: an fMRI study in severe major depressive disorder. Biol Psychiatry. 2008 Feb 15;63(4):369-76. doi: 10.1016/j.biopsych.2007.05.033. Epub 2007 Sep 21. PMID 17888408
- [Background] Moses-Kolko EL, Perlman SB, Wisner KL, James J, Saul AT, Phillips ML. Abnormally reduced dorsomedial prefrontal cortical activity and effective connectivity with amygdala in response to negative emotional faces in postpartum depression. Am J Psychiatry. 2010 Nov;167(11):1373-80. doi: 10.1176/appi.ajp.2010.09081235. Epub 2010 Sep 15. PMID 20843875
- [Background] Moses-Kolko EL, Fraser D, Wisner KL, James JA, Saul AT, Fiez JA, Phillips ML. Rapid habituation of ventral striatal response to reward receipt in postpartum depression. Biol Psychiatry. 2011 Aug 15;70(4):395-9. doi: 10.1016/j.biopsych.2011.02.021. Epub 2011 Apr 20. PMID 21507385
- [Background] Epstein J, Pan H, Kocsis JH, Yang Y, Butler T, Chusid J, Hochberg H, Murrough J, Strohmayer E, Stern E, Silbersweig DA. Lack of ventral striatal response to positive stimuli in depressed versus normal subjects. Am J Psychiatry. 2006 Oct;163(10):1784-90. doi: 10.1176/ajp.2006.163.10.1784. PMID 17012690
- [Background] Smoski MJ, Felder J, Bizzell J, Green SR, Ernst M, Lynch TR, Dichter GS. fMRI of alterations in reward selection, anticipation, and feedback in major depressive disorder. J Affect Disord. 2009 Nov;118(1-3):69-78. doi: 10.1016/j.jad.2009.01.034. Epub 2009 Mar 3. PMID 19261334
- [Background] Hamilton JP, Gotlib IH. Neural substrates of increased memory sensitivity for negative stimuli in major depression. Biol Psychiatry. 2008 Jun 15;63(12):1155-62. doi: 10.1016/j.biopsych.2007.12.015. Epub 2008 Feb 20. PMID 18281017
- [Background] Schmidt PJ, Nieman LK, Danaceau MA, Adams LF, Rubinow DR. Differential behavioral effects of gonadal steroids in women with and in those without premenstrual syndrome. N Engl J Med. 1998 Jan 22;338(4):209-16. doi: 10.1056/NEJM199801223380401. PMID 9435325
- [Background] Roca CA, Schmidt PJ, Deuster PA, Danaceau MA, Altemus M, Putnam K, Chrousos GP, Nieman LK, Rubinow DR. Sex-related differences in stimulated hypothalamic-pituitary-adrenal axis during induced gonadal suppression. J Clin Endocrinol Metab. 2005 Jul;90(7):4224-31. doi: 10.1210/jc.2004-2525. Epub 2005 May 10. PMID 15886244
- [Background] Leibenluft E, Schmidt PJ, Turner EH, Danaceau MA, Ashman SB, Wehr TA, Rubinow DR. Effects of leuprolide-induced hypogonadism and testosterone replacement on sleep, melatonin, and prolactin secretion in men. J Clin Endocrinol Metab. 1997 Oct;82(10):3203-7. doi: 10.1210/jcem.82.10.4270. PMID 9329339
- [Background] Bloch M, Rotenberg N, Koren D, Klein E. Risk factors associated with the development of postpartum mood disorders. J Affect Disord. 2005 Sep;88(1):9-18. doi: 10.1016/j.jad.2005.04.007. PMID 15979150
- [Background] Berman KF, Schmidt PJ, Rubinow DR, Danaceau MA, Van Horn JD, Esposito G, Ostrem JL, Weinberger DR. Modulation of cognition-specific cortical activity by gonadal steroids: a positron-emission tomography study in women. Proc Natl Acad Sci U S A. 1997 Aug 5;94(16):8836-41. doi: 10.1073/pnas.94.16.8836. PMID 9238064
- [Background] Schmidt PJ, Steinberg EM, Negro PP, Haq N, Gibson C, Rubinow DR. Pharmacologically induced hypogonadism and sexual function in healthy young women and men. Neuropsychopharmacology. 2009 Feb;34(3):565-76. doi: 10.1038/npp.2008.24. Epub 2008 Mar 19. PMID 18354393
- [Background] Le Strat Y, Dubertret C, Le Foll B. Prevalence and correlates of major depressive episode in pregnant and postpartum women in the United States. J Affect Disord. 2011 Dec;135(1-3):128-38. doi: 10.1016/j.jad.2011.07.004. Epub 2011 Jul 29. PMID 21802737
- [Background] Vesga-Lopez O, Schneier FR, Wang S, Heimberg RG, Liu SM, Hasin DS, Blanco C. Gender differences in generalized anxiety disorder: results from the National Epidemiologic Survey on Alcohol and Related Conditions (NESARC). J Clin Psychiatry. 2008 Oct;69(10):1606-16. Epub 2008 Sep 23. PMID 19192444
- [Background] Steingold KA, Matt DW, DeZiegler D, Sealey JE, Fratkin M, Reznikov S. Comparison of transdermal to oral estradiol administration on hormonal and hepatic parameters in women with premature ovarian failure. J Clin Endocrinol Metab. 1991 Aug;73(2):275-80. doi: 10.1210/jcem-73-2-275. PMID 1906893
- [Background] Chetkowski RJ, Meldrum DR, Steingold KA, Randle D, Lu JK, Eggena P, Hershman JM, Alkjaersig NK, Fletcher AP, Judd HL. Biologic effects of transdermal estradiol. N Engl J Med. 1986 Jun 19;314(25):1615-20. doi: 10.1056/NEJM198606193142505. PMID 3012339
- [Background] Rice VC, Richard-Davis G, Saleh AA, Ginsburg KA, Mammen EF, Moghissi K, Leach R. Fibrinolytic parameters in women undergoing ovulation induction. Am J Obstet Gynecol. 1993 Dec;169(6):1549-53. doi: 10.1016/0002-9378(93)90434-k. PMID 8267060
- [Background] Saleh AA, Ginsburg KA, Duchon TA, Dorey LG, Hirata J, Alshameeri RS, Dombrowski MP, Mammen EF. Hormonal contraception and platelet function. Thromb Res. 1995 May 15;78(4):363-7. doi: 10.1016/0049-3848(95)91464-v. PMID 7631316
- [Background] Sulak PJ, Cressman BE, Waldrop E, Holleman S, Kuehl TJ. Extending the duration of active oral contraceptive pills to manage hormone withdrawal symptoms. Obstet Gynecol. 1997 Feb;89(2):179-83. doi: 10.1016/S0029-7844(96)00488-7. PMID 9015017
- [Background] Feuillan PP, Jones JV, Barnes KM, Oerter-Klein K, Cutler GB Jr. Boys with precocious puberty due to hypothalamic hamartoma: reproductive axis after discontinuation of gonadotropin-releasing hormone analog therapy. J Clin Endocrinol Metab. 2000 Nov;85(11):4036-8. doi: 10.1210/jcem.85.11.6951. PMID 11095429
- [Background] Feuillan PP, Jones JV, Barnes K, Oerter-Klein K, Cutler GB Jr. Reproductive axis after discontinuation of gonadotropin-releasing hormone analog treatment of girls with precocious puberty: long term follow-up comparing girls with hypothalamic hamartoma to those with idiopathic precocious puberty. J Clin Endocrinol Metab. 1999 Jan;84(1):44-9. doi: 10.1210/jcem.84.1.5409. PMID 9920060
- [Background] Gambrell RD Jr. The role of hormones in the etiology and prevention of endometrial cancer. Clin Obstet Gynaecol. 1986 Dec;13(4):695-723. PMID 3791826
- [Background] Nieman, L. K. & Loriaux, D. L. Estrogens and progestins. in Textbook of pharmacology 695-716 (W.B. Saunders Company, 1992).
- [Background] Jick H, Derby LE, Myers MW, Vasilakis C, Newton KM. Risk of hospital admission for idiopathic venous thromboembolism among users of postmenopausal oestrogens. Lancet. 1996 Oct 12;348(9033):981-3. doi: 10.1016/S0140-6736(96)07114-0. PMID 8855853
- [Background] Daly E, Vessey MP, Hawkins MM, Carson JL, Gough P, Marsh S. Risk of venous thromboembolism in users of hormone replacement therapy. Lancet. 1996 Oct 12;348(9033):977-80. doi: 10.1016/S0140-6736(96)07113-9. PMID 8855852
- [Background] Grodstein F, Stampfer MJ, Goldhaber SZ, Manson JE, Colditz GA, Speizer FE, Willett WC, Hennekens CH. Prospective study of exogenous hormones and risk of pulmonary embolism in women. Lancet. 1996 Oct 12;348(9033):983-7. doi: 10.1016/S0140-6736(96)07308-4. PMID 8855854
- [Background] Cushman M, Kuller LH, Prentice R, Rodabough RJ, Psaty BM, Stafford RS, Sidney S, Rosendaal FR; Women's Health Initiative Investigators. Estrogen plus progestin and risk of venous thrombosis. JAMA. 2004 Oct 6;292(13):1573-80. doi: 10.1001/jama.292.13.1573. PMID 15467059
- [Background] Stampfer MJ, Colditz GA, Willett WC, Manson JE, Rosner B, Speizer FE, Hennekens CH. Postmenopausal estrogen therapy and cardiovascular disease. Ten-year follow-up from the nurses' health study. N Engl J Med. 1991 Sep 12;325(11):756-62. doi: 10.1056/NEJM199109123251102. PMID 1870648
- [Background] Wassertheil-Smoller S, Hendrix SL, Limacher M, Heiss G, Kooperberg C, Baird A, Kotchen T, Curb JD, Black H, Rossouw JE, Aragaki A, Safford M, Stein E, Laowattana S, Mysiw WJ; WHI Investigators. Effect of estrogen plus progestin on stroke in postmenopausal women: the Women's Health Initiative: a randomized trial. JAMA. 2003 May 28;289(20):2673-84. doi: 10.1001/jama.289.20.2673. PMID 12771114
- [Background] Mandel FP, Geola FL, Meldrum DR, Lu JH, Eggena P, Sambhi MP, Hershman JM, Judd HL. Biological effects of various doses of vaginally administered conjugated equine estrogens in postmenopausal women. J Clin Endocrinol Metab. 1983 Jul;57(1):133-9. doi: 10.1210/jcem-57-1-133. PMID 6304131
- [Background] Melis GB, Fruzzetti F, Paoletti AM, Carmassi F, Fioretti P. Fibrinopeptide A plasma levels during low-estrogen oral contraceptive treatment. Contraception. 1984 Dec;30(6):575-83. doi: 10.1016/0010-7824(84)90007-6. PMID 6241562
- [Background] Barrett-Connor E, Bush TL. Estrogen and coronary heart disease in women. JAMA. 1991 Apr 10;265(14):1861-7. PMID 2005736
- [Background] Manson JE, Hsia J, Johnson KC, Rossouw JE, Assaf AR, Lasser NL, Trevisan M, Black HR, Heckbert SR, Detrano R, Strickland OL, Wong ND, Crouse JR, Stein E, Cushman M; Women's Health Initiative Investigators. Estrogen plus progestin and the risk of coronary heart disease. N Engl J Med. 2003 Aug 7;349(6):523-34. doi: 10.1056/NEJMoa030808. PMID 12904517
- [Background] Willett WC, Manson JE, Grodstein F, Stampfer MJ, Colditz GA. Re: "combined postmenopausal hormone therapy and cardiovascular disease: toward resolving the discrepancy between observational studies and the women's health initiative clinical trial". Am J Epidemiol. 2006 Jun 1;163(11):1067-8; author reply 1068-9. doi: 10.1093/aje/kwj156. Epub 2006 Apr 26. No abstract available. PMID 16641306
- [Background] Prentice RL, Langer RD, Stefanick ML, Howard BV, Pettinger M, Anderson GL, Barad D, Curb JD, Kotchen J, Kuller L, Limacher M, Wactawski-Wende J; Women's Health Initiative Investigators. Combined analysis of Women's Health Initiative observational and clinical trial data on postmenopausal hormone treatment and cardiovascular disease. Am J Epidemiol. 2006 Apr 1;163(7):589-99. doi: 10.1093/aje/kwj079. Epub 2006 Feb 16. PMID 16484450
- [Background] Grodstein F, Manson JE, Stampfer MJ. Hormone therapy and coronary heart disease: the role of time since menopause and age at hormone initiation. J Womens Health (Larchmt). 2006 Jan-Feb;15(1):35-44. doi: 10.1089/jwh.2006.15.35. PMID 16417416
- [Background] Prentice RL, Langer R, Stefanick ML, Howard BV, Pettinger M, Anderson G, Barad D, Curb JD, Kotchen J, Kuller L, Limacher M, Wactawski-Wende J; Women's Health Initiative Investigators. Combined postmenopausal hormone therapy and cardiovascular disease: toward resolving the discrepancy between observational studies and the Women's Health Initiative clinical trial. Am J Epidemiol. 2005 Sep 1;162(5):404-14. doi: 10.1093/aje/kwi223. Epub 2005 Jul 20. PMID 16033876
- [Background] Lobo RA. Evaluation of cardiovascular event rates with hormone therapy in healthy, early postmenopausal women: results from 2 large clinical trials. Arch Intern Med. 2004 Mar 8;164(5):482-4. doi: 10.1001/archinte.164.5.482. No abstract available. PMID 15006823
- [Background] Hsia J, Langer RD, Manson JE, Kuller L, Johnson KC, Hendrix SL, Pettinger M, Heckbert SR, Greep N, Crawford S, Eaton CB, Kostis JB, Caralis P, Prentice R; Women's Health Initiative Investigators. Conjugated equine estrogens and coronary heart disease: the Women's Health Initiative. Arch Intern Med. 2006 Feb 13;166(3):357-65. doi: 10.1001/archinte.166.3.357. PMID 16476878
- [Background] Cirillo DJ, Wallace RB, Rodabough RJ, Greenland P, LaCroix AZ, Limacher MC, Larson JC. Effect of estrogen therapy on gallbladder disease. JAMA. 2005 Jan 19;293(3):330-9. doi: 10.1001/jama.293.3.330. PMID 15657326
- [Background] Petitti DB, Sidney S, Perlman JA. Increased risk of cholecystectomy in users of supplemental estrogen. Gastroenterology. 1988 Jan;94(1):91-5. doi: 10.1016/0016-5085(88)90614-2. PMID 3335303
- [Background] Steinauer JE, Waetjen LE, Vittinghoff E, Subak LL, Hulley SB, Grady D, Lin F, Brown JS. Postmenopausal hormone therapy: does it cause incontinence? Obstet Gynecol. 2005 Nov;106(5 Pt 1):940-5. doi: 10.1097/01.AOG.0000180394.08406.15. PMID 16260510
- [Background] Grodstein F, Lifford K, Resnick NM, Curhan GC. Postmenopausal hormone therapy and risk of developing urinary incontinence. Obstet Gynecol. 2004 Feb;103(2):254-60. doi: 10.1097/01.AOG.0000107290.33034.6f. PMID 14754692
- [Background] Hendrix SL, Cochrane BB, Nygaard IE, Handa VL, Barnabei VM, Iglesia C, Aragaki A, Naughton MJ, Wallace RB, McNeeley SG. Effects of estrogen with and without progestin on urinary incontinence. JAMA. 2005 Feb 23;293(8):935-48. doi: 10.1001/jama.293.8.935. PMID 15728164
- [Background] Wingo PA, Layde PM, Lee NC, Rubin G, Ory HW. The risk of breast cancer in postmenopausal women who have used estrogen replacement therapy. JAMA. 1987 Jan 9;257(2):209-15. PMID 3795407
- [Background] Grady, D. & Ernster, V. Invited Commentary: Does Postmenopausal Hormone Therapy Cause Breast Cancer? Am. J. Epidemiol. 134, 1396-1400 (1991).
- [Background] Colditz GA, Hankinson SE, Hunter DJ, Willett WC, Manson JE, Stampfer MJ, Hennekens C, Rosner B, Speizer FE. The use of estrogens and progestins and the risk of breast cancer in postmenopausal women. N Engl J Med. 1995 Jun 15;332(24):1589-93. doi: 10.1056/NEJM199506153322401. PMID 7753136
- [Background] Breast cancer and hormone replacement therapy: collaborative reanalysis of data from 51 epidemiological studies of 52,705 women with breast cancer and 108,411 women without breast cancer. Collaborative Group on Hormonal Factors in Breast Cancer. Lancet. 1997 Oct 11;350(9084):1047-59. PMID 10213546
- [Background] Chen WY, Manson JE, Hankinson SE, Rosner B, Holmes MD, Willett WC, Colditz GA. Unopposed estrogen therapy and the risk of invasive breast cancer. Arch Intern Med. 2006 May 8;166(9):1027-32. doi: 10.1001/archinte.166.9.1027. PMID 16682578
- [Background] Stefanick ML, Anderson GL, Margolis KL, Hendrix SL, Rodabough RJ, Paskett ED, Lane DS, Hubbell FA, Assaf AR, Sarto GE, Schenken RS, Yasmeen S, Lessin L, Chlebowski RT; WHI Investigators. Effects of conjugated equine estrogens on breast cancer and mammography screening in postmenopausal women with hysterectomy. JAMA. 2006 Apr 12;295(14):1647-57. doi: 10.1001/jama.295.14.1647. PMID 16609086
- [Background] Chlebowski RT, Hendrix SL, Langer RD, Stefanick ML, Gass M, Lane D, Rodabough RJ, Gilligan MA, Cyr MG, Thomson CA, Khandekar J, Petrovitch H, McTiernan A; WHI Investigators. Influence of estrogen plus progestin on breast cancer and mammography in healthy postmenopausal women: the Women's Health Initiative Randomized Trial. JAMA. 2003 Jun 25;289(24):3243-53. doi: 10.1001/jama.289.24.3243. PMID 12824205
- [Background] Gann PH, Morrow M. Combined hormone therapy and breast cancer: a single-edged sword. JAMA. 2003 Jun 25;289(24):3304-6. doi: 10.1001/jama.289.24.3304. No abstract available. PMID 12824214
- [Background] Li CI, Malone KE, Porter PL, Weiss NS, Tang MT, Cushing-Haugen KL, Daling JR. Relationship between long durations and different regimens of hormone therapy and risk of breast cancer. JAMA. 2003 Jun 25;289(24):3254-63. doi: 10.1001/jama.289.24.3254. PMID 12824206
- [Background] Sturmer T, Manson JE. Estrogens and breast cancer: does timing really matter? J Clin Epidemiol. 2004 Aug;57(8):763-5. doi: 10.1016/j.jclinepi.2003.12.018. No abstract available. PMID 15485726
- [Background] Rossouw JE, Anderson GL, Prentice RL, LaCroix AZ, Kooperberg C, Stefanick ML, Jackson RD, Beresford SA, Howard BV, Johnson KC, Kotchen JM, Ockene J; Writing Group for the Women's Health Initiative Investigators. Risks and benefits of estrogen plus progestin in healthy postmenopausal women: principal results From the Women's Health Initiative randomized controlled trial. JAMA. 2002 Jul 17;288(3):321-33. doi: 10.1001/jama.288.3.321. PMID 12117397
- [Background] Henzel, M. R. Contraceptive hormones and their clinical use. in Reproductive endocrinology: physiology, pathophysiology and clinical management 643-682 (W.B. Saunders Company, 1986).
- [Background] Hommer RE, Meyer A, Stoddard J, Connolly ME, Mogg K, Bradley BP, Pine DS, Leibenluft E, Brotman MA. Attention bias to threat faces in severe mood dysregulation. Depress Anxiety. 2014 Jul;31(7):559-65. doi: 10.1002/da.22145. Epub 2013 Jun 24. PMID 23798350

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hormone Sensitive Women (HS+) | Hormone Insensitive Women (HS-)
Started | 13 | 10
Completed | 13 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hormone Sensitive Women (HS+) | Hormone Insensitive Women (HS-) | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.81 (6.46) | 37.15 (2.82) | 35.77 (5.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Mean Threat Processing Bias During Visual Dot-probe Paradigm Over Time
Description: This outcome measure determines the extent to which irritability is characterized by dysfunctional threat processing during reproductive hormone challenge relative to baseline in HS+ and HS- by examining threat attention bias assessed during the visual dot-probe paradigm.
  The Visual Dot-Probe Paradigm asks participants to detect a target stimulus that is embedded in a matrix of distracting stimuli (e.g., a target stimulus, an angry face, might be embedded in a matrix of neutral distractor faces). Attention biases are inferred from faster response times to detect a threatening stimulus in a matrix of neutral stimuli relative to response time to detect neutral stimuli in neutral matrices. Thus, positive times reflect attention bias toward threat, whereas negative times reflect attention bias away from threat.
Time Frame: up to 6 weeks
Population: All available data are reported. Data are missing for participants who had insufficient time to complete the task or due to computer malfunction.
Measure: Mean (Standard Deviation); unit: attention bias in milliseconds
Groups:
- Hormone Sensitive Women (HS+): Participants will take leuprolide acetate (lupron) via intramuscular injection, for 2 months. Participants will take 2 mg of estradiol twice daily and 200 mg of progesterone twice daily for 2 weeks.
  Leuprolide Acetate 3.75 MG/ML: 3.75 mg/month leuprolide acetate intramuscular injection
  Estradiol 2 Mg tablet: 2 mg estradiol tablet
  Micronized progesterone: 200 mg micronized progesterone tablets
  Hormone sensitive women were those who experienced at least a 30% increase in negative mood symptoms as defined by the IDAS during hormone addback.
- Hormone Insensitive Women (HS-): Participants will take leuprolide acetate (lupron) via intramuscular injection, for 2 months. Participants will take 2 mg of estradiol twice daily and 200 mg of progesterone twice daily for 2 weeks.
  Leuprolide Acetate 3.75 MG/ML: 3.75 mg/month leuprolide acetate intramuscular injection
  Estradiol 2 Mg tablet: 2 mg estradiol tablet
  Micronized progesterone: 200 mg micronized progesterone tablets
  Hormone Insensitive women did not experience a 30% increase in negative mood symptoms during hormone addback.
Arm/Group | Hormone Sensitive Women (HS+) | Hormone Insensitive Women (HS-)
Number analyzed (Participants) | 10 | 9
attention bias in milliseconds
  Baseline (Visit 3) | -0.57 (18.92) | 36.92 (110.98)
  Hormone Addback (Visit 6) | -9.04 (31.57) | -42.35 (102.99)
Statistical Analysis 1: Comparison: Hormone Sensitive Women (HS+) vs Hormone Insensitive Women (HS-); Test type: Superiority; p = 0.160, repeated measures ANOVA; F statistic = 2.164

2. Primary Outcome: Mean Right Amygdala-medial Prefrontal Cortex BOLD Connectivity During Implicit Emotion Face Processing Task Over Time
Description: This outcome measure determines the extent to which irritability is characterized by dysfunctional threat processing during reproductive hormone challenge relative to baseline in HS+ and HS-. By examining amygdala-medial prefrontal cortex (PFC) Blood-oxygen-level-dependent (BOLD) connectivity in response to threatening faces on the implicit emotion face processing fMRI task in HS+ (compared with HS-) during hormone challenge relative to baseline.
  The implicit emotion face processing task asks participants to identify the gender of angry, happy, and fearful faces at 50%, 100% and 150% emotion intensity presented in random order for 2000 milliseconds followed by jittered fixation. Trials appear in 3 blocks, generating 30 trials of each emotion at each intensity and 90 neutral face emotion trials.
Time Frame: up to 6 weeks
Population: Participants exceeding the motion threshold and those completing the task incorrectly were excluded.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Hormone Sensitive Women (HS+) | Hormone Insensitive Women (HS-)
Number analyzed (Participants) | 11 | 6
arbitrary units
  Baseline (Visit 3) | 0.0174 (0.0606) | 0.0533 (0.0338)
  Hormone Addback (Visit 6) | -0.0114 (0.0751) | 0.00804 (0.0943)
Statistical Analysis 1: Comparison: Hormone Sensitive Women (HS+) vs Hormone Insensitive Women (HS-); Test type: Superiority; p = 0.1922, ANOVA; F statistic = 1.74

3. Primary Outcome: Mean Left Amygdala-medial Prefrontal Cortex BOLD Connectivity During Implicit Emotion Face Processing Task Over Time
Description: This outcome measure determines the extent to which irritability is characterized by dysfunctional threat processing during reproductive hormone challenge relative to baseline in HS+ and HS-. By examining amygdala-medial prefrontal cortex (PFC) connectivity in response to threatening faces on the implicit emotion face processing fMRI task in HS+ (compared with HS-) during hormone challenge relative to baseline.
  The implicit emotion face processing task asks participants to identify the gender of angry, happy, and fearful faces at 50%, 100% and 150% emotion intensity presented in random order for 2000 milliseconds followed by jittered fixation. Trials appear in 3 blocks, generating 30 trials of each emotion at each intensity and 90 neutral face emotion trials.
Time Frame: up to 6 weeks
Population: Participants exceeding the motion threshold and those completing the task incorrectly were excluded.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Hormone Sensitive Women (HS+) | Hormone Insensitive Women (HS-)
Number analyzed (Participants) | 11 | 6
arbitrary units
  Baseline (Visit 3) | 0.0247 (0.0653) | 0.0213 (0.0374)
  Hormone Addback (Visit 6) | -0.0192 (0.0893) | 0.00111 (0.0884)
Statistical Analysis 1: Comparison: Hormone Sensitive Women (HS+) vs Hormone Insensitive Women (HS-); Test type: Superiority; p = 0.368, ANOVA; F statistic = 0.837

4. Primary Outcome: Mean Reactive Aggression During Hormone Addback Over Time
Description: This outcome measure determines the extent to which HS+ is characterized by reactive aggression during hormone addback relative to baseline in the target population. Reactive aggression will be defined as the number of point subtractions the participant makes during the Point Subtraction Aggression Paradigm.
  Point Subtraction Aggression Paradigm measures relational aggression (approach behavior) in response to frustration. In the task, participants are asked to press a button to accrue money or press another button to subtract money from a (fictional) partner at no direct gain to themselves. Frustration is induced by periodic subtractions of their own money, which is attributed to the partner.
Time Frame: up to 6 weeks
Measure: Mean (Standard Deviation); unit: Number of subtraction responses
Arm/Group | Hormone Sensitive Women (HS+) | Hormone Insensitive Women (HS-)
Number analyzed (Participants) | 13 | 10
Number of subtraction responses
  Baseline (Visit 3) | 103.08 (121.68) | 129.20 (105.76)
  Hormone Addback (Visit 6) | 34.62 (44.84) | 54.90 (71.85)
Statistical Analysis 1: Comparison: Hormone Sensitive Women (HS+) vs Hormone Insensitive Women (HS-); Test type: Superiority; p = 0.881, ANOVA; F statistic = 0.23

5. Primary Outcome: Mean BOLD Activation of the Right Amygdala During the Affective Posner Task Over Time
Description: This outcome measure determines the extent to which HS+ is characterized by BOLD activation of the right amygdala in response to frustrative non-reward (FNR) in the Affective Posner Task during hormone addback relative to baseline in the target population.
  The Affective Posner Task tests whether HS+ is characterized by reduced subcortical activation in response to frustration. This task is divided into 3 runs: during Run 1 (practice run), participants receive accurate feedback about their performance on the task and do not win or lose money; during Run 2, participants receive accurate feedback about their performance and win or lose 50 cents per trial; and during Run 3 (frustration), participants are told they must respond accurately to win money, but participants are given feedback that they responded too slowly on 60% of accurate trials, regardless of their performance.
Time Frame: up to 6 weeks
Population: Participants exceeding the motion threshold were excluded as were those with signal loss.
Measure: Mean (Standard Deviation); unit: Arbitrary Units
Arm/Group | Hormone Sensitive Women (HS+) | Hormone Insensitive Women (HS-)
Number analyzed (Participants) | 11 | 9
Arbitrary Units
  Baseline (Visit 3) | -0.04544 (0.100148) | 0.037334 (0.137479)
  Hormone Addback (Visit 6) | 0.022654 (0.071363) | -0.15643 (0.089792)
Statistical Analysis 1: Comparison: Hormone Sensitive Women (HS+) vs Hormone Insensitive Women (HS-); Test type: Superiority; p = 0.000723, ANOVA; F statistic = 16.541

6. Primary Outcome: Mean BOLD Activation of the Left Amygdala During the Affective Posner Task Over Time
Description: This outcome measure determines the extent to which HS+ is characterized by BOLD activation of the left amygdala in response to frustrative non-reward (FNR) in the Affective Posner Task during hormone addback relative to baseline in the target population.
  The Affective Posner Task tests whether HS+ is characterized by reduced subcortical activation in response to frustration. This task is divided into 3 runs: during Run 1 (practice run), participants receive accurate feedback about their performance on the task and do not win or lose money; during Run 2, participants receive accurate feedback about their performance and win or lose 50 cents per trial; and during Run 3 (frustration), participants are told they must respond accurately to win money, but participants are given feedback that they responded too slowly on 60% of accurate trials, regardless of their performance.
Time Frame: up to 6 weeks
Population: Participants exceeding the motion threshold were excluded.
Measure: Mean (Standard Deviation); unit: Arbitrary Units
Arm/Group | Hormone Sensitive Women (HS+) | Hormone Insensitive Women (HS-)
Number analyzed (Participants) | 12 | 9
Arbitrary Units
  Baseline (Visit 3) | 0.005316917 (0.10109272) | -0.009866667 (0.12208237)
  Hormone Addback (Visit 6) | -0.047401917 (0.19032614) | -0.086876444 (0.11792679)
Statistical Analysis 1: Comparison: Hormone Sensitive Women (HS+) vs Hormone Insensitive Women (HS-); Test type: Superiority; p = 0.791, ANOVA; F statistic = 0.072

7. Primary Outcome: Mean BOLD Activation of the Right Caudate During the Affective Posner Task Over Time
Description: This outcome measure determines the extent to which HS+ is characterized by BOLD activation of the right caudate in response to frustrative non-reward (FNR) in the Affective Posner Task during hormone addback relative to baseline in the target population.
  The Affective Posner Task tests whether HS+ is characterized by reduced subcortical activation in response to frustration. This task is divided into 3 runs: during Run 1 (practice run), participants receive accurate feedback about their performance on the task and do not win or lose money; during Run 2, participants receive accurate feedback about their performance and win or lose 50 cents per trial; and during Run 3 (frustration), participants are told they must respond accurately to win money, but participants are given feedback that they responded too slowly on 60% of accurate trials, regardless of their performance.
Time Frame: up to 6 weeks
Measure: Mean (Standard Deviation); unit: Arbitrary Units
Arm/Group | Hormone Sensitive Women (HS+) | Hormone Insensitive Women (HS-)
Number analyzed (Participants) | 13 | 10
Arbitrary Units
  Baseline (Visit 3) | -0.069919077 (0.11155759) | 0.061407 (0.15720728)
  Hormone Addback (Visit 6) | 0.045146154 (0.1320315) | 0.0058011 (0.15927022)
Statistical Analysis 1: Comparison: Hormone Sensitive Women (HS+) vs Hormone Insensitive Women (HS-); Test type: Superiority; p = 0.0372, ANOVA; F statistic = 4.952

8. Primary Outcome: Mean BOLD Activation of the Left Caudate During the Affective Posner Task Over Time
Description: This outcome measure determines the extent to which HS+ is characterized by BOLD activation of the left caudate in response to frustrative non-reward (FNR) in the Affective Posner Task during hormone addback relative to baseline in the target population.
  The Affective Posner Task tests whether HS+ is characterized by reduced subcortical activation in response to frustration. This task is divided into 3 runs: during Run 1 (practice run), participants receive accurate feedback about their performance on the task and do not win or lose money; during Run 2, participants receive accurate feedback about their performance and win or lose 50 cents per trial; and during Run 3 (frustration), participants are told they must respond accurately to win money, but participants are given feedback that they responded too slowly on 60% of accurate trials, regardless of their performance.
Time Frame: up to 6 weeks
Population: Participants with signal loss were excluded.
Measure: Mean (Standard Deviation); unit: Arbitrary Units
Arm/Group | Hormone Sensitive Women (HS+) | Hormone Insensitive Women (HS-)
Number analyzed (Participants) | 12 | 10
Arbitrary Units
  Baseline (Visit 3) | -0.043943333 (0.19455199) | 0.0077258 (0.18794868)
  Hormone Addback (Visit 6) | 0.059099917 (0.09144575) | -0.049988 (0.17179757)
Statistical Analysis 1: Comparison: Hormone Sensitive Women (HS+) vs Hormone Insensitive Women (HS-); Test type: Superiority; p = 0.0861, ANOVA; F statistic = 3.258

9. Primary Outcome: Mean BOLD Activation of the Right Putamen During the Affective Posner Task Over Time
Description: This outcome measure determines the extent to which HS+ is characterized by BOLD activation of the right putamen in response to frustrative non-reward (FNR) in the Affective Posner Task during hormone addback relative to baseline in the target population.
  The Affective Posner Task tests whether HS+ is characterized by reduced subcortical activation in response to frustration. This task is divided into 3 runs: during Run 1 (practice run), participants receive accurate feedback about their performance on the task and do not win or lose money; during Run 2, participants receive accurate feedback about their performance and win or lose 50 cents per trial; and during Run 3 (frustration), participants are told they must respond accurately to win money, but participants are given feedback that they responded too slowly on 60% of accurate trials, regardless of their performance.
Time Frame: up to 6 weeks
Population: Participants with signal loss were excluded.
Measure: Mean (Standard Deviation); unit: Arbitrary Units
Arm/Group | Hormone Sensitive Women (HS+) | Hormone Insensitive Women (HS-)
Number analyzed (Participants) | 13 | 9
Arbitrary Units
  Baseline (Visit 3) | -0.007560692 (0.09339182) | 0.002542222 (0.17117375)
  Hormone Addback (Visit 6) | 0.036225385 (0.1357793) | -0.080736333 (0.08070693)
Statistical Analysis 1: Comparison: Hormone Sensitive Women (HS+) vs Hormone Insensitive Women (HS-); Test type: Superiority; p = 0.139, ANOVA; F statistic = 2.370

10. Primary Outcome: Mean BOLD Activation of the Left Putamen During the Affective Posner Task Over Time
Description: This outcome measure determines the extent to which HS+ is characterized by BOLD activation of the left putamen in response to frustrative non-reward (FNR) in the Affective Posner Task during hormone addback relative to baseline in the target population.
  The Affective Posner Task tests whether HS+ is characterized by reduced subcortical activation in response to frustration. This task is divided into 3 runs: during Run 1 (practice run), participants receive accurate feedback about their performance on the task and do not win or lose money; during Run 2, participants receive accurate feedback about their performance and win or lose 50 cents per trial; and during Run 3 (frustration), participants are told they must respond accurately to win money, but participants are given feedback that they responded too slowly on 60% of accurate trials, regardless of their performance.
Time Frame: up to 6 weeks
Measure: Mean (Standard Deviation); unit: Arbitrary Units
Arm/Group | Hormone Sensitive Women (HS+) | Hormone Insensitive Women (HS-)
Number analyzed (Participants) | 13 | 10
Arbitrary Units
  Baseline (Visit 3) | -0.001223462 (0.11938667) | 0.0383029 (0.2004158)
  Hormone Addback (Visit 6) | 0.048155385 (0.13830948) | -0.021029 (0.17785651)
Statistical Analysis 1: Comparison: Hormone Sensitive Women (HS+) vs Hormone Insensitive Women (HS-); Test type: Superiority; p = 0.237, ANOVA; F statistic = 1.484

11. Primary Outcome: Mean BOLD Activation of the Right Nucleus Accumbens During the Affective Posner Task Over Time
Description: This outcome measure determines the extent to which HS+ is characterized by BOLD activation of the right nucleus accumbens in response to frustrative non-reward (FNR) in the Affective Posner Task during hormone addback relative to baseline in the target population.
  The Affective Posner Task tests whether HS+ is characterized by reduced subcortical activation in response to frustration. This task is divided into 3 runs: during Run 1 (practice run), participants receive accurate feedback about their performance on the task and do not win or lose money; during Run 2, participants receive accurate feedback about their performance and win or lose 50 cents per trial; and during Run 3 (frustration), participants are told they must respond accurately to win money, but participants are given feedback that they responded too slowly on 60% of accurate trials, regardless of their performance.
Time Frame: up to 6 weeks
Population: Participants with signal loss were excluded.
Measure: Mean (Standard Deviation); unit: Arbitrary Units
Arm/Group | Hormone Sensitive Women (HS+) | Hormone Insensitive Women (HS-)
Number analyzed (Participants) | 12 | 9
Arbitrary Units
  Baseline (Visit 3) | 0.044384167 (0.17318851) | 0.052685333 (0.13130308)
  Hormone Addback (Visit 6) | -0.005181667 (0.16825616) | -0.006394444 (0.21780392)
Statistical Analysis 1: Comparison: Hormone Sensitive Women (HS+) vs Hormone Insensitive Women (HS-); Test type: Superiority; p = 0.910, ANOVA; F statistic = 0.013

12. Primary Outcome: Mean BOLD Activation of the Left Nucleus Accumbens During the Affective Posner Task Over Time
Description: This outcome measure determines the extent to which HS+ is characterized by BOLD activation of the left nucleus accumbens in response to frustrative non-reward (FNR) in the Affective Posner Task during hormone addback relative to baseline in the target population.
  The Affective Posner Task tests whether HS+ is characterized by reduced subcortical activation in response to frustration. This task is divided into 3 runs: during Run 1 (practice run), participants receive accurate feedback about their performance on the task and do not win or lose money; during Run 2, participants receive accurate feedback about their performance and win or lose 50 cents per trial; and during Run 3 (frustration), participants are told they must respond accurately to win money, but participants are given feedback that they responded too slowly on 60% of accurate trials, regardless of their performance.
Time Frame: up to 6 weeks
Population: Participants with signal loss were excluded.
Measure: Mean (Standard Deviation); unit: Arbitrary Units
Arm/Group | Hormone Sensitive Women (HS+) | Hormone Insensitive Women (HS-)
Number analyzed (Participants) | 11 | 10
Arbitrary Units
  Baseline (Visit 3) | -0.028451818 (0.13242342) | 0.0691907 (0.24951478)
  Hormone Addback (Visit 6) | 0.031632727 (0.25999277) | -0.072512 (0.16302971)
Statistical Analysis 1: Comparison: Hormone Sensitive Women (HS+) vs Hormone Insensitive Women (HS-); Test type: Superiority; p = 0.0449, ANOVA; F statistic = 4.609

13. Secondary Outcome: Correlation Between the Inventory of Depressive and Anxiety Symptoms (IDAS) Ill -0.8Scale and Threat Attention Bias
Description: This outcome measure determines the extent to which irritability is characterized by dysfunctional reward processing during reproductive hormone challenge in HS+ and HS- by examining the correlation between the Inventory of Depressive and Anxiety Symptoms (IDAS) Ill Temper (i.e., irritability) Scale and threat attention bias.
Time Frame: Endpoint (week 6)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Hormone Sensitive Women (HS+) | Hormone Insensitive Women (HS-)
Number analyzed (Participants) | 10 | 9
correlation coefficient | -0.35 [-0.8 to 0.36] | 0.11 [-0.6 to 0.72]
Statistical Analysis 1: Comparison: Hormone Sensitive Women (HS+); Test type: Superiority; p = 0.322, Pearson's Correlation Coefficient
Statistical Analysis 2: Comparison: Hormone Insensitive Women (HS-); Test type: Superiority; p = 0.772, Pearson's Correlation Coefficient

14. Secondary Outcome: Correlation Between the Inventory of Depressive and Anxiety Symptoms (IDAS) Ill Temper Scale and Right Amygdala-medial Prefrontal Cortex (PFC) BOLD Connectivity.
Description: This outcome measure determines the extent to which irritability is characterized by dysfunctional reward processing during reproductive hormone challenge in HS+ and HS- by examining the correlation between the IDAS Ill Temper (i.e., irritability) Scale and amygdala-medial PFC connectivity in HS+.
Time Frame: Endpoint (week 6)
Population: Participants exceeding the motion threshold and those completing the task incorrectly were excluded.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Hormone Sensitive Women (HS+) | Hormone Insensitive Women (HS-)
Number analyzed (Participants) | 11 | 6
correlation coefficient | -0.57 [-0.87 to 0.05] | -0.08 [-0.84 to 0.78]
Statistical Analysis 1: Comparison: Hormone Sensitive Women (HS+); Test type: Superiority; p = 0.068, Pearson correlation; Pearson's r = -0.5683140
Statistical Analysis 2: Comparison: Hormone Insensitive Women (HS-); Test type: Superiority; p = 0.8759289, Pearson correlation; Pearson's r = -0.0829040

15. Secondary Outcome: Correlation Between the Inventory of Depressive and Anxiety Symptoms (IDAS) Ill Temper Scale and Left Amygdala-medial Prefrontal Cortex (PFC) BOLD Connectivity.
Description: as for outcome 14
Time Frame: Endpoint (week 6)
Population: Participants exceeding the motion threshold and those completing the task incorrectly were excluded.
Measure: Mean (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Hormone Sensitive Women (HS+) | Hormone Insensitive Women (HS-)
Number analyzed (Participants) | 11 | 6
correlation coefficient | -0.13 [-0.68 to 0.51] | 0.49 [-0.53 to 0.93]
Statistical Analysis 1: Comparison: Hormone Sensitive Women (HS+); Test type: Superiority; p = 0.70859639, Pearson correlation; Pearson's r = -0.1275539
Statistical Analysis 2: Comparison: Hormone Insensitive Women (HS-); Test type: Superiority; p = 0.2617744, Pearson correlation; Pearson's r = 0.49225646

16. Secondary Outcome: Correlation Between Irritability and Reactive Aggression During Hormone Addback
Description: This outcome measure determines the degree of irritability and reactive aggression in HS+ during hormone addback and its relationship to the target population. Irritability will be defined as score on the IDAS Ill Temper Scale. Reactive aggression will be defined as the number of point subtractions the participant makes during the Point Subtraction Aggression Paradigm.
  The Point Subtraction Aggression Paradigm measures relational aggression (approach behavior) in response to frustration. In the task, participants are asked to press a button to ac
Time Frame: Endpoint (week 6)
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Hormone Sensitive Women (HS+) | Hormone Insensitive Women (HS-)
Number analyzed (Participants) | 13 | 10
correlation coefficient | 0.18 [-0.42 to 0.66] | 0.03 [-0.61 to 0.65]
Statistical Analysis 1: Comparison: Hormone Sensitive Women (HS+); Test type: Superiority; p = 0.568, Pearson's Correlation Coefficient
Statistical Analysis 2: Comparison: Hormone Insensitive Women (HS-); Test type: Superiority; p = 0.944, Pearson's Correlation Coefficient

17. Secondary Outcome: Correlation Between Irritability Subcortical Activation in HS+ During Hormone Addback
Description: This outcome measure determines the degree of subcortical (amygdala, caudate, putamen, and nucleus accumbens) activation in HS+ during hormone addback and it's relationship to the target population. The activation in amygdala and ventral striatum (caudate, putamen, nucleus accumbens) regions of interest (ROIs) will be assessed during the Affective Posner Task.
  The Affective Posner Task tests whether HS+ is characterized by reduced subcortical activation in response to frustration. This task is divided into 3 runs: during Run 1 (practice run), participants receive accurate feedback about their performance on the task and do not win or lose money; during Run 2, participants receive accurate feedback about their performance and win or lose 50 cents per trial; and during Run 3 (frustration), participants are told they must respond accurately to win money, but participants are given feedback that they responded too slowly on 60% of accurate trials, regardless of their performance.
Time Frame: Endpoint (week 6)
Population: The a priori hypothesis focused on the HS+ group only.
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Arm/Group | Hormone Sensitive Women (HS+) | Hormone Insensitive Women (HS-)
Number analyzed (Participants) | 13 | 0
correlation coefficient | 0.47 [-0.11 to 0.81] |
Statistical Analysis 1: Comparison: Hormone Sensitive Women (HS+); Test type: Superiority; p = 0.103, Pearson's Correlation Coefficient

ADVERSE EVENTS:
Time Frame: From Study visit 3 (intervention start) through visit 7 (Follow-Up), a total of approximately 9 weeks.
Arm/Group | Hormone Sensitive Women (HS+) | Hormone Insensitive Women (HS-)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/10
Other Adverse Events (participants affected / at risk) | 12/13 | 9/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hormone Sensitive Women (HS+) (N=13) | Hormone Insensitive Women (HS-) (N=10)
Bloating (Gastrointestinal disorders) | 3 (3) | 3 (3)
Low back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
General musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0)
Cramps (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Headache (General disorders) | 7 (7) | 4 (4)
Migraine (Vascular disorders) | 2 (2) | 1 (1)
Occular migraine (Vascular disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 8 (9) | 4 (5)
Arm soreness (Lupron IM injection) (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Arm soreness (COVID vaccine IM injection) (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Hot flashes (Reproductive system and breast disorders) | 9 (10) | 8 (8)
Fever (COVID-19 infection) (Infections and infestations) | 1 (1) | 0 (0)
Anosmia (COVID-19 infection) (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 Infection (Infections and infestations) | 1 (1) | 0 (0)
Dry cough (Seasonal allergies) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Gastrointestinal upset (Gastrointestinal disorders) | 3 (3) | 4 (4)
Mood swings (Psychiatric disorders) | 1 (1) | 0 (0)
Spotting (Reproductive system and breast disorders) | 6 (6) | 2 (2)
Intrusive thoughts (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (5) | 3 (3)
Anhedonia (Psychiatric disorders) | 2 (2) | 0 (0)
Depressed mood (Psychiatric disorders) | 2 (2) | 0 (0)
Irritability (Psychiatric disorders) | 4 (4) | 3 (3)
Low libido (Psychiatric disorders) | 1 (1) | 0 (0)
Weight gain (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Early insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Late insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Breast tenderness (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 6 (7) | 1 (1)
Difficulty concentrating (Psychiatric disorders) | 1 (1) | 0 (0)
Emotional sensitivity (Psychiatric disorders) | 4 (4) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hematoma (IM injection) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Yeast infection (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hormonal acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hair loss (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cervical mucus (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fever (Infections and infestations) | 0 (0) | 1 (1)
Hip pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Frequent urination (Renal and urinary disorders) | 0 (0) | 1 (1)
Vivid dreams (Psychiatric disorders) | 0 (0) | 1 (1)
Passive suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/20/NCT04051320/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-05): https://cdn.clinicaltrials.gov/large-docs/20/NCT04051320/ICF_001.pdf